CLINICAL TRIAL: NCT05972616
Title: A Single-center Review of the Performance of Induce Biologics NMP™ in Patients Who Have Undergone Interbody Fusion for Degenerative Disease of the Lumbar Spine
Brief Title: Natural Matrix Protein™ (NMP™) in Interbody Lumbar Fusion
Status: Completed | Type: Observational
Sponsor: Induce Biologics USA Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SIL-2023-NMP
Record Dates: First submitted 2023-07-12; First posted 2023-08-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Degenerative Disc Disease
Keywords: lumbar spine fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMP: Have clinical or radiological evidence of degenerative disc disease of the lumbar spine.
  Have been treated with NMP™ during a lumbar spinal fusion procedure.
  Interventions: Biological: Natural Matrix Protein (NMP)

INTERVENTIONS:
Biological: Natural Matrix Protein (NMP) — human bone allograft

SUMMARY:
The objective of this study is to evaluate the performance of Induce Biologics NMP™ when used to promote interbody fusion for degenerative disease of the lumbar spine.

DETAILED DESCRIPTION:
The study involves a retrospective review of patients' medical records and prospective collection of CT scans, X-rays, and patient centered outcome questionnaires.

The study population will include up to 135 patients of the Spine Institute of Louisiana (SIL) who have been treated with Induce Biologics NMP™ during a lumbar interbody fusion. All subjects who meet all inclusion criteria and do not meet any exclusion criteria will be included in the study.

There will be a single Prospective Visit in this study. This visit will be scheduled at the 12-month (± 2 mo) post-surgery time point.

ELIGIBILITY:
Inclusion Criteria:

1. Have clinical or radiological evidence of degenerative disc disease of the lumbar spine.
2. Have been treated with Induce Biologics NMP™ during a lumbar spinal fusion procedure.
3. Be at least 18 years of age.
4. Have current contact information.
5. Be willing and able to provide written Informed Consent for the prospective part of study participation.
6. Be willing and able to undergo a CT-scan and X-rays.
7. Be willing and able to complete patient centered outcome questionnaires.

Exclusion Criteria:

1. Currently imprisoned.
2. Currently experiencing major mental illness (psychosis, schizophrenia, major affective disorder) which in the opinion of the investigator may indicate that the symptoms are psychological rather than of physical origin.
3. X-rays or CT-scan are contraindicated.
4. Any previous lumbar fusion or arthroplasty surgery at the index level(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 135 patients of the Spine Institute of Louisiana (SIL) who have been treated with Induce Biologics NMP™ during a lumbar interbody fusion. All subjects who meet all inclusion criteria and do not meet any exclusion criteria will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Radiographic fusion rate | 12-months post-surgery
  CT scans will be graded from 0 (no boney ingrowth) to 3 (complete bridging) and A (no evidence of supplemental fixation failure) or B (evidence of supplemental fixation failure).
  Fusion will be defined as a CT grade of 3A with less than 3 degrees of motion at the index level on flexion and extension x-rays.

SECONDARY OUTCOMES:
Change in disability score assessed by Oswestry Disability Index | Baseline to 12 months post-operative
  Disability will be assessed using the Oswestry Disability Index (ODI). ODI is a questionnaire to collect a patient's responses to questions about perceived function (disability) in 10 everyday activities in patients with acute or chronic low back pain. Each question consists of 6 statements about 1 activity which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest. The scores are combined to a single score from 0 (no disability) to 50 (completely disabled)
Change in disability score assessed by the 12-Item Short Form Survey version 2 | Baseline to 12 months post-operative
  Disability will be assessed by the 12-Item Short Form Survey version 2 (SF-12v2).
  The SF-12 is is a questionnaire to collect a patient's responses to 12 questions about their physical and mental health. It is often used as a quality of life measure. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The minimum score for MCS-12 is 3.2 and the maximum score is 77.9. The minimum score for PCS-12 is 9.9 and the maximum score 76.0. The lower the score the worse the health.
Change in pain score - for the Back | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for back pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks. The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced.
Change in pain score - for the Left Leg | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for left leg pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced.
Change in pain score - for the Right Leg | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for right leg pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks. The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced.
Adverse Events (AE) related to NMP | Baseline to 12 months post-operative
  All Adverse Events (AE) will be documented in detail and followed to a satisfactory resolution regardless of the cause. The intensity of the adverse event is determined by the investigator using the following definitions:
  Mild: The AE is commonly asymptomatic or causes minimal symptoms and does not require any active intervention.
  Moderate: The AE causes discomfort and requires treatment but does not pose any significant or permanent risk to harm the subject. It may or may not require any intervention.
  Severe: Incapacitating with inability to perform usual activities. It is a definite hazard to health, reduced life expectancy, death, or life threatening, necessitates medical or surgical intervention to preclude permanent disability.
  The number of mild, moderate and severe AE determined to be related to NMP™ will be collected and reported.
Change in neurologic status | Baseline to 12 months post-operative
  Neurologic status will be assessed using a grading scale during a physical exam. The patient will be scored by a clinician as to motor strength (0 to 5 paralysis to normal), sensory function based on response to touch and pin prick (0 absent, 1 numbness, 2 normal, 3 hypersensitive) and reflexes (0 absent, 1 diminished, 2 normal, 3 hyperactive, 4 hyperactive with clonus).
Revisions/reoperations | Baseline to 12 months post-operative
  number of revisions or reoperations performed will be collected and reported.
Duration of hospitalization | time of surgery to time of discharge, assessed up to 12 months
  number of days in hospital post-operation will be collected and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Nunley, MD, Principal Investigator — Spine Institute of Louisiana
Locations (1):
- Spine Institute of Louisiana, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No